CLINICAL TRIAL: NCT04414072
Title: Effect of Bariatric Surgery
Brief Title: Local GIT Hormones After Bariatric Maneuvers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Amr Abdel Hameed El heny, Assistant professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 367177
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: surgeries
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- laparoscopic sleeve gastrectomy (Active Comparator)
  Interventions: Procedure: sleeve gastrectomy with loop bipartition
- mini gastric bypass (Active Comparator)
  Interventions: Procedure: sleeve gastrectomy with loop bipartition
- sleeve gastrectomy with loop bipartition (Active Comparator)
  Interventions: Procedure: sleeve gastrectomy with loop bipartition

INTERVENTIONS:
Procedure: sleeve gastrectomy with loop bipartition — operations to decrease weight
  Other Names: minigastric bypass

SUMMARY:
Background: Many of the beneficial metabolic effects of bariatric surgery have been attributed to altered peptide hormone profiles, especially involving pancreatic and gut peptides.

Objectives: assess the effects of bariatric procedures (sleeve gastrectomy, minigastric bypass and sleeve gastrectomy with loop bipartition) on GIT hormones. Methods: Prospective randomized study which was carried out in the department of General Surgery, Minia University hospital during the period from February 2018 to February 2019. This study included 3 groups subjected to different operations; each group consisted of 50 patients.

DETAILED DESCRIPTION:
Prospective randomized study which was carried out in the department of General Surgery, Minia University hospital during the period from February 2018 to February 2019. This study included 3 groups subjected to different operations; each group consisted of 50 patients. Age ranging from 20 to 50 years old and body weight ranging from 100 to 200 Kg, and subjected to laparoscopic sleeve gastrectomy, mini gastric bypass and sleeve gastrectomy with loop bipartition. Each patient was thoroughly evaluated by a multidisciplinary team (Nutritionist, Endocrinologist, Psychologist, and Surgeon) using a standardized protocol. Follow up was done after two weeks and after 2 months.

ELIGIBILITY:
Inclusion Criteria:

All morbid obese patients

-

Exclusion Criteria:

GIT diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
hormonal change | one year
  GIT hormones (Ghrelin, secretin, PYY, GLP-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code